CLINICAL TRIAL: NCT06347068
Title: Study of Administration of T Cells Expressing B7-H3 Specific Chimeric Antigen Receptors and Containing the Inducible Caspase 9 Safety Switch in Subjects With Triple Negative Breast Cancer
Brief Title: Study of Autologous CAR-T Cells Targeting B7-H3 in TNBC iC9-CAR.B7-H3 T Cells
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2128-ATL; P50CA058223-29A1 (NIH)
Record Dates: First submitted 2024-03-22; First posted 2024-04-04 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Relapse; Resistant Cancer; Triple Negative Breast Cancer
Keywords: cellular therapy; biologic therapy
MeSH Terms: conditions — Breast Neoplasms; Recurrence; Triple Negative Breast Neoplasms | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- iC9-CAR.B7-H3 T cells (Experimental): Specimen will be collected to prepare the iC9-CAR.B7-H3 T cells. Disease-fighting T cells will be isolated and modified to prepare the iC9-CAR.B7-H3 T cells. In part 2, the iC9-CAR.B7-H3 T cells are given by infusion after completion of lymphodepletion chemotherapy.
  Interventions: Biological: iC9-CAR.B7-H3 T Cell Therapy; Drug: cyclophosphamide; Drug: fludarabine

INTERVENTIONS:
Biological: iC9-CAR.B7-H3 T Cell Therapy — iC9-CAR.B7-H3 T cells will then be administered intravenously
  Other Names: iC9-CAR.B7-H3 T cells
Drug: cyclophosphamide — cyclophosphamide 300 mg/m2 IV will be given.
  Other Names: Cytoxan
Drug: fludarabine — fludarabine 30 mg/m2 IV will be given.
  Other Names: Fludara; Fludarabine Phosphate

SUMMARY:
This phase 1, single-center, open-label study explores the safety of escalating doses of chimeric antigen receptor T cells (CAR-T) cells in subjects with relapsed/refractory triple-negative breast cancer (TNBC).

DETAILED DESCRIPTION:
T lymphocyte chimeric antigen receptor cells against the B7-H3 antigen (iC9-CAR.B7-H3 T cells) treatment is experimental and has not been approved by the Food and Drug Administration. The safety of iC9-CAR.B7-H3 T cells will be investigated using a modified 3+3 design. The data from the dose escalation will be used to determine a recommended phase 2 dose (RP2D), which will be decided based on the maximum tolerated dose (MTD) and additional factors such as the ability to manufacture sufficient cells for infusion.

Subjects with TNBC who meet procurement eligibility criteria will have cells collected to manufacture iC9-CAR.B7-H3 T cells. Eligible subjects will receive lymphodepletion with cyclophosphamide and fludarabine.

ELIGIBILITY:
Inclusion Criteria:

Unless otherwise noted, subjects must meet all of the following criteria to participate in in all phases of the study:

1. Written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization for release of personal health information explained to, understood by and signed by the subject or legally authorized representative.
2. Age ≥ 18 years at the time of consent.
3. Karnofsky score of > 60% (see APPENDIX VI- Karnofsky Scale))
4. Histologically confirmed TNBC (ER-, PR-, HER2-negative)

   1. ER- and PR-negative: defined as < 1% staining by immunohistochemistry (IHC)
   2. HER2-negative: defined as IHC 0-1+ or fluorescence in situ hybridization (FISH) ratio < 2.0

Exclusion Criteria:

1. Patients with a history of symptomatic CNS involvement or multiple metastases requiring whole-brain radiation.
2. Subjects with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
3. Subject does not have a measurable and or evaluable disease as defined by RECIST 1.1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Toxicity: NCI-CTCAE | Up to 4 weeks
  Toxicity will be graded as the Number of participants with adverse events (AE)s
  AEs will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.
Toxicity: Cytokine Release Syndrome (CRS) | Up to 8 weeks after infusion of Biological/Vaccine
  CRS will be graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) CRS Consensus Grading. Grade 1 - Mild: Fever ≥38^ o C, No hypotension, No hypoxia, Grade 2 - Moderate: Fever ≥38^ o C, Hypotension not requiring vasopressors, Hypoxia requiring low-flow nasal cannula (≤6 L/minute) or blow-by, Grade 3 - Severe: Fever ≥ 38^ o C, Hypotension requiring a vasopressor with or without vasopressin, Hypoxia requiring high-flow nasal cannula (>6 L/minute), facemask, nonrebreather mask, or Venturi mask, Grade 4 - Life-threatening: Fever ≥38^oC, Hypotension requiring multiple vasopressors (excluding vasopressin), Hypoxia requiring positive pressure (e.g. Continuous positive airway pressure, BiPAP, intubation, mechanical ventilation), Grade 5 - Death
Toxicity: Immune effector cell-associated neurotoxicity syndrome (ICANS) | Up to 4 weeks
  Neurotoxicity will be graded according to the Immune effector cell-associated neurotoxicity syndrome (ICANS) criteria.
  Immune effector cell-associated neurotoxicity syndrome (ICANS) symptoms will be graded according to the criteria outlined in the protocol on a scale from 1 (mild) to 4 (critical). Cytokine release syndrome (CRS) will be graded according to criteria outlined in the protocol on a scale from 1 (mild) to grade 5 (death).

SECONDARY OUTCOMES:
The recommended phase 2 dose (RP2D) NCI-CTCAE v5. | Up to 4 weeks
  The RP2D of iC9-CAR.B7-H3 T cells will be determined based on modified 3+3 dose finding rules and the tolerability of iC9-CAR.B7-H3 T cells will be assessed by NCI-CTCAE v5 criteria.
The recommended phase 2 dose (RP2D) CRS Grading | Up to 4 weeks
  The RP2D of iC9-CAR.B7-H3 T cells will be determined based on modified 3+3 dose finding rules and the tolerability of iC9-CAR.B7-H3 T cells will be assessed byASTCT Consensus CRS Grading Criteria.
The recommended phase 2 dose (RP2D) | Up to 4 weeks
  The RP2D of iC9-CAR.B7-H3 T cells will be determined based on modified 3+3 dose finding rules and the tolerability of iC9-CAR.B7-H3 T cells will be assessed by ASTCT Consensus ICANS Grading Criteria.
Objective response rate | Up to 2 years
  Objective response rate is defined as the percentage of subjects achieving a confirmed partial response (PR) or better (≥ PR) based on RECIST 1.1 criteria.
  Complete response - Disappearance of all target lesions. Any pathological lymph node (LN) must be <10mm. Partial response: At least a 30% decrease in the sum of the largest distance (LD) of the target lesions. Progressive Disease (PD): At least a 20% increase in the sum of the LD of the target lesions taking as reference the smallest sum LD recorded since the treatment started including baseline if that is the smallest in the study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. The appearance of one or more new lesions also constitutes PD. Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD since the treatment started.
Progression Free Survival (PFS) | Up to 2 years
  PFS will be measured from the first day of lymphodepletion chemotherapy prior to iC9-CAR.B7-H3 T cell infusion to progression per RECIST 1.1 or death.
Overall Survival (OS) | Up to 2 years
  OS will be measured from the first day of lymphodepleting chemotherapy prior to iC9-CAR.B7-H3 T cell infusion to the date of death for any cause.
Duration of Response (DOR) | Up to 2 years
  DOR is defined as the time from documentation of PR or better to progressive disease (PD) based on RECIST 1.1 and/or irRECIST.
  Per immune-related Response Evaluation Criteria in Solid Tumors (irRECIST) for target and/or non-target lesions and assessed by imaging: Complete Response (irCR), Disappearance of all lesions, no new lesions, lymph nodes < 10 mm in short axis; Partial Response (irPR), ≥30% decrease in the sum of target lesions and non-target lesions are irNN; Stable response (irSD), not meeting criteria for irCR, irPR, or irPD; Progressive Disease (irPD), ≥20% increase in tumor burden and minimum 5 mm absolute increase in compared to nadir; for no new non-target or (irNN) and where irPR or irPD are confirmed by a repeat, consecutive assessment no less than 4 weeks later.

CONTACTS AND LOCATIONS:
Overall Officials: Yara E Abdou, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials